CLINICAL TRIAL: NCT04954976
Title: Epidemiologic Study of Orthodontic Retention Practices in France
Brief Title: Orthodontic Retention In France - ORIF
Acronym: ORIF
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AL - RNI ORIF
Record Dates: First submitted 2021-06-16; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Orthodontic Retention Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Orthodontic retention procedures survey — The survey was composed of eight parts, about sociodemographic status, retention system selection, choice of fixed and removable retention system, retention period, supervision, given instruction and needs for practice guidelines.

SUMMARY:
The goal of this study is to survey retention procedures used by French orthodontists, and evaluate the needs for practice guidelines. The hypothesis is that there is no consensus among orthodontists, requiring practice homogenization via expert guidelines. Similar studies have been driven in others European countries (such as Swiss, the Netherlands, Lithuania and Norway), but not in France.

DETAILED DESCRIPTION:
Questionnaire aggregating 27 questions on orthodontic retention strategies, was sent to a professional list of French orthodontists from health authorities. The survey was composed of eight parts, about sociodemographic status, retention system selection, choice of fixed and removable retention system, retention period, supervision, given instruction and needs for practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* All French Specialist orthodontists trained in France who answer the survey

Exclusion Criteria:

* Non-specialist orthodontists, not trained in France

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French orthodontists
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Description of technics | Day0 = Response to the Suvey
  Retention system selection, choice of fixed and removable retention system, retention period, supervision, given instruction and needs for practice guidelines.
Description of materials | Day0 = Response to the Suvey
  Retention system selection, choice of fixed and removable retention system, retention period, supervision, given instruction and needs for practice guidelines.
Description of retention strategies used by clinicians. | Day0 = Response to the Suvey
  Retention system selection, choice of fixed and removable retention system, retention period, supervision, given instruction and needs for practice guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No
No IPD